CLINICAL TRIAL: NCT05930561
Title: A Phase 2 Randomized, Active-Controlled, Double-masked Trial of Intravitreal 4D-150 Gene Therapy in Adults With Diabetic Macular Edema (SPECTRA)
Brief Title: 4D-150 in Patients With Diabetic Macular Edema
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4D-150-C002
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: Retinal gene therapy; Intravitreal gene therapy; DME; SPECTRA
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: In Dose Confirmation (Part 1), subjects (n=12-18) will be sequentially assigned to one of two open-label dose levels of 4D-150 (n=6-9 per dose level). In Dose Expansion (Part 2), subjects (n=54) will be randomized to receive one of two dose levels of 4D-150 (n=18 per dose level) based on results from Dose Confirmation, or aflibercept control (n=18). Subjects will be masked to treatment arm in Dose Expansion (Part 2).
Who Masked: Participant, Outcomes Assessor
Masking Description: No masking in Dose Confirmation (Part 1). In Dose Expansion (Part 2), participants and outcomes assessors will be masked to the treatment arm for the duration of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 4D-150 Part 1 Dose Confirmation Dose Level 1 (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Part 1 Dose Confirmation Dose Level 2 (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Part 2 Dose Expansion Dose Level 1 (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Part 2 Dose Expansion Dose Level 2 (Experimental): 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1.
  Interventions: Biological: 4D-150 IVT
- 4D-150 Part 2 Dose Expansion Control (Active Comparator): Aflibercept at a fixed regimen will be administered.
  Interventions: Biological: Aflibercept IVT

INTERVENTIONS:
Biological: 4D-150 IVT — 4D-150: AAV-based gene therapy comprised of miRNA targeting VEGF-C and codon-optimized sequence encoding aflibercept.
  Arms: 4D-150 Part 1 Dose Confirmation Dose Level 1; 4D-150 Part 1 Dose Confirmation Dose Level 2; 4D-150 Part 2 Dose Expansion Dose Level 1; 4D-150 Part 2 Dose Expansion Dose Level 2
Biological: Aflibercept IVT — Commercially available Active Comparator
  Other Names: Eylea
  Arms: 4D-150 Part 2 Dose Expansion Control

SUMMARY:
Phase 2 randomized, active-controlled, double-masked, dose-ranging trial in adults with Diabetic Macular Edema (DME).

DETAILED DESCRIPTION:
This Phase 2 trial is a prospective, multicenter, randomized, active-controlled, double-masked dose-ranging trial to evaluate the safety and efficacy of 4D-150 in adults with DME. The trial will be conducted in two parts: Dose Confirmation and Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Type I or Type II diabetes mellitus with macular thickening secondary to DME involving the center of the fovea; diagnosis of DME must be within 2 years of Screening
* CST ≥ 350 μm (Spectralis SD-OCT) in the study eye at Screening, confirmed by the independent reading center
* Demonstrate clinical response to on-study aflibercept injection in the study eye.
* Decreased visual acuity attributable primarily to DME
* BCVA in the study eye between 25 and 83 ETDRS letters, inclusive (~20/320 and 20/25, respectively) at Screening
* Study eye amenable to IVT injection
* Sufficient clear ocular media, pupil dilation and fixation in the study eye to permit adequate imaging; ability to perform tests of visual and retinal function and structure; and ability to comply with other protocol-specified procedures
* Provide written informed consent

Exclusion Criteria:

* Macular edema in the study eye considered to be secondary to a cause other than DME
* Systemic anti-VEGF treatment (e.g. sunitinib, bevacizumab, pazopanib) within 6 months, or anticipated need for systemic anti-VEGF therapy during study participation
* Systemic corticosteroids (oral, intravenous, intramuscular, intra-articular) or other immunosuppressive medications within 3 months
* Received an investigational drug, agent, device, or therapy (ocular or non-ocular) in the 3 months (or at least 5 half-lives, whichever is longer) prior to 4D-150 administration (Day 1)
* Prior gene therapy (ocular or non-ocular) and/or ocular stem cell therapy in either eye
* Any concurrent ocular condition in the study eye that is likely to require surgical intervention (e.g. cataract surgery) during the 2 year (104 week) study duration

Note: Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of TEAEs and SAEs, including clinically significant changes in safety parameters (Part 1) | 60 months
Annualized number of aflibercept injections in the study eye (Part 2) | 52 weeks

SECONDARY OUTCOMES:
Mean cumulative number of aflibercept injections over time | 52 weeks
Change from baseline in BCVA as assessed using the ETDRS Visual Acuity Chart at Weeks 52 and 104 | 104 weeks
Change from baseline in CST measured by spectral domain optical coherence tomography (SD-OCT) at Weeks 104 | 104 weeks

OTHER OUTCOMES:
Incidence and severity of treatment-emergent adverse events and serious adverse events, including clinically significant changes in safety parameters | 104 weeks
Development of anti-drug antibodies to capsid protein (4D-R100) and the transgene product (aflibercept) and change in antibody titers in subjects receiving 4D-150 | 104 weeks
Change in levels of aflibercept protein in aqueous humor and serum overtime | 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julie Clark, MD, Study Director — 4D Molecular Therapeutics
Locations (6):
- United States (5):
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Verum Research, LLC, Eugene, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Austin Clinical Research, Austin, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
- Emanuelli Research and Development Center, Arecibo, Puerto Rico